CLINICAL TRIAL: NCT06730581
Title: Phase II Clinical Trial of Utidelone Capsule in the Treatment of Advanced Solid Tumor Patients
Brief Title: Utidelone Capsule Monotherapy for Patients with Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2403
Record Dates: First submitted 2024-11-21; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer Adenocarcinoma Metastatic; Ovarian Cancer; Bile Duct Cancer
Keywords: Gastric Cancer; Ovarian Cancer; bile duct cancer
MeSH Terms: conditions — Ovarian Neoplasms; Bile Duct Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gastric cancer group (Experimental)
  Interventions: Drug: Utidelone Capsule 60mg/m2/d
- Ovarian and cholangiocarcinoma groups (Experimental)
  Interventions: Drug: Utidelone capsule 75mg/m2
- Other oncology indications (including esophageal cancer, liver cancer, colorectal cancer, cervical c (Experimental)
  Interventions: Drug: Utidelone Capsule

INTERVENTIONS:
Drug: Utidelone Capsule 60mg/m2/d — 60mg/m2/d, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Gastric cancer group
Drug: Utidelone capsule 75mg/m2 — 75mg/m2/d, D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Ovarian and cholangiocarcinoma groups
Drug: Utidelone Capsule — Dosing regimens were determined based on the results of gastric and ovarian cancer dosing regimens.D1-D5 for 5 consecutive days, every 21 days as a treatment cycle.
  Arms: Other oncology indications (including esophageal cancer, liver cancer, colorectal cancer, cervical c

SUMMARY:
This trial is an open, multicenter, phase II clinical trial to evaluate the efficacy and safety of Utidelone capsules in patients with advanced solid tumors. The target population of the study is patients with advanced solid tumors (gastric cancer, ovarian cancer, cholangiocarcinoma and other tumors (esophageal cancer, hepatocellular carcinoma, colorectal cancer, cervical cancer). The number of evaluable cases for tumor enrollment in gastric, ovarian, and bile duct cancers will be 20 cases each, and the total number of other tumors (including esophageal, liver, colorectal, and cervical cancers) will be no more than 40 cases. Patients who met the enrollment criteria received Utidelone capsule (UTD2) monotherapy.

ELIGIBILITY:
Inclusion Criteria:

-

1、 For participants with advanced gastric cancer:Histologically and/or cytologically confirmed unresectable HER2-negative locally advanced or recurrent/metastatic gastric or gastroesophageal junction adenocarcinoma (according to the 2019 WHO Classification of Digestive System Oncology).

2、 For participants with advanced cholangiocarcinoma:Histologically and/or cytologically, patients were diagnosed with surgically unresectable advanced or metastatic cholangiocarcinoma.

3、 For participants with advanced ovarian cancer:A histologically or pathologically confirmed diagnosis of high-grade serous ovarian cancer was consistent with platinum-resistant recurrent ovarian cancer (progression within 6 months after the last platinum-based chemotherapy) according to the 2020 WHO histopathological classification of ovarian tumors.

4、 For participants with other tumors:

1. Esophageal cancer: locally advanced recurrent or metastatic squamous esophageal cancer confirmed by histology or cytology.
2. Hepatocellular carcinoma: clinically diagnosed or histologically/cytologically confirmed diagnosis of inoperable resectable or metastatic hepatocellular carcinoma (HCC) (according to the Guidelines for the Management of Primary Hepatocellular Carcinoma (2024 edition)); Child-Pugh score ≤ 7.
3. Colorectal cancer: unresectable advanced/metastatic colorectal cancer (mCRC) confirmed by histology or cytology.
4. Recurrent or metastatic cervical cancer confirmed by histopathology, not amenable to radical surgical resection and/or radical radiotherapy, and pathologic type of squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.

5、For all participants:

1. Subjects must give informed consent to the study prior to the study, and voluntarily sign a written informed consent form (ICF), understanding and agreeing to comply with the study requirements and test procedures;
2. ≥18 years old and ≤70 years old;
3. According to RECIST v1.1, patients had at least one target lesion (non-radiotherapy field) that could be measured by computed tomography (CT) or magnetic resonance imaging (MRI) (longest diameter ≥10mm, lymph node diameter ≥15mm, scan layer thickness ≤ 5mm).
4. Have received at least one standard systemic therapy, and the number of previous systemic anti-tumor therapy lines is ≤4 (neoadjuvant and adjuvant chemotherapy regiments are not considered prior systemic therapy unless disease progression occurs during their chemotherapy or within 6 months after the last chemotherapy);
5. The blood routine examination within 1 week before enrollment was basically normal (the normal value of the laboratory of each research center was the standard); No rhG-CSF, blood transfusion /EPO and other drugs were used within 14 days before enrollment.

   a. White blood cell count (WBC) ≥3.5 × 109/L b.Neutrophil count (ANC) ≥ 1.5 × 109/L; c.Platelet count (PLT) ≥ 100 × 109/L; d.Hemoglobin ≥ 9.0 g/dL.
6. Within one week before enrollment, the blood biochemistry test was basically normal (based on the normal values of each research center laboratory):

   a.Total bilirubin (TBIL) ≤ 1.5 x Upper limit of normal value (ULN) b.SGPT/ALT ≤ 3 × ULN (liver metastasis patients ≤ 5 × ULN); c.SGOT/AST ≤ 3 × ULN (liver metastasis patients ≤ 5 × ULN); d.The creatinine clearance rate (Ccr) is ≥ 60 ml/min (Cockcroft Gault formula).
7. adequate coagulation function, defined as INR or PT ≤1.5 times ULN; If the subject was receiving anticoagulant therapy, as long as the PT was within the prescribed range of anticoagulant drugs.
8. ECOG 0-1 with an expected survival of more than 12 weeks;
9. Patients of childbearing potential had to consent to use a reliable contraceptive method (hormonal or barrier methods or abstinence) with their partner simultaneously during the trial and for at least 3 months after the last dose; Female patients of reproductive age had to have a negative blood or urine pregnancy test before enrollment.

Exclusion Criteria:

-

1、 For participants with advanced gastric cancer:Patients with HER2-positive disease.

2、 For participants with advanced ovarian cancer: 1) Having a clear cell, mucinous or sarcomatous histology, containing mixed tumours of any histological type, or low grade/borderline ovarian cancer; 2) Platinum-refractory ovarian cancer: tumor progression assessed within 1 month after the last dose of platinum therapy.

3、 For all participants:

1. Other malignancies within 5 years, excluding cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary carcinoma of the thyroid;
2. Received nitrosourea or mitomycin C within 6 weeks prior to the first use of the study drug; Anti-tumor therapy, including chemotherapy, radiotherapy, biotargeted therapy, immunotherapy, etc. within 4 weeks or 5 half-lives (whichever is shorter) prior to the first use of the investigational drug; Oral fluorouracil, small molecule targeted drugs, or endocrine therapy within 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug, whichever is shorter; Use of traditional Chinese medicine or proprietary Chinese medicine with anti-tumor indications within 2 weeks prior to the first use of the investigational drug.
3. had major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first use of the study drug, or required elective surgery during the trial period.
4. Patients with peripheral neuropathy CTCAE 5.0 grade ≥2.
5. The adverse reactions of previous antineoplastic therapy have not recovered to CTCAE 5.0 grade ≤1 (except for toxicities without safety risk judged by investigators, such as alopecia).
6. Patients who had previously used Utidelone injection.
7. Patients with gastrointestinal bleeding, active gastrointestinal ulcers or gastrointestinal obstruction (including paralytic ileus), gastrointestinal perforation or fistula, and intraperitoneal abscesses within 6 months prior to the first use of the investigational drug;
8. Patients with dysphagia, or other factors that affect the oral administration and absorption of drugs, or who require parenteral nutrition;
9. Clinically active brain metastases, spinal cord compression, or spread of pia meningioma, defined as symptomatic or requiring steroid hormone or anticonvulsant therapy to control related symptoms; Patients with confirmed progression of brain metastases within 2 months after radiotherapy or other local treatment;
10. Clinically severe lung injury caused by concurrent lung disease, including but not limited to any underlying lung disease (i.e., pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion, etc., with clinical symptoms requiring intervention within 3 months prior to the first use of the investigational drug);
11. Patients with clinical symptoms of cancerous ascites, pleural effusion and pericardial effusion requiring puncture and drainage; Or had undergone drainage of ascites, pleural effusion, or pericardial effusion within 30 days prior to the first use of the study drug.
12. Imaging shows that the tumor has invaded the vicinity of important blood vessels or the investigator determines that the patient's tumor is highly likely to invade important blood vessels during treatment and cause fatal massive bleeding;
13. Have a history of severe cardiovascular and cerebrovascular disease, including but not limited to:

    1. Have severe heart rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree Ⅱ-Ⅲ atrioventricular block, etc.; At rest, QTcF> 450 ms in men or 470ms in women was examined by 12-lead electrocardiogram (Fredericia's formula, see Appendix IV);
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular event within 6 months prior to first use of the study drug;
    3. Clinically uncontrollable hypertension;
    4. Other researchers have identified a high risk of heart disease.
14. Patients with uncontrolled diabetes within 3 months prior to first use of the study drug.
15. Patients with active hepatitis B and/or hepatitis C, i.e. HBsAg positive and/or HBcAb positive with HBV DNA positive and/or anti-HCV positive and HCV RNA positive; Positive for human immunodeficiency virus (HIV) antibodies; The specific antibody of treponema pallidum was positive.
16. Those who have an active infection and currently require systemic anti-infective therapy.
17. Had an active autoimmune disease that required systemic treatment (i.e., disease modulators, corticosteroids, or immunosuppressive drugs) within 2 years prior to enrollment. Replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered a systemic treatment.
18. Women who are pregnant or nursing or plan to become pregnant during the study period.
19. Patients with mental disorders or poor compliance.
20. Known allergy to the investigational drug or any of its excipients.
21. Concurrent participation in another interventional clinical trial or use of another investigational treatment.
22. The researchers believe that the subjects have a history of serious systemic disease, or other reasons should not be enrolled in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR）according to the RECIST 1.1. | 18 months

SECONDARY OUTCOMES:
Progression-Free Survival, PFS | 18 months
Clinical Benefit Rate （CBR）according to the RECIST 1.1. | 18 months
CA125 versus baseline remission rate, only the ovarian cancer group was eligible | 18 months
Maximum (or peak) serum concentration-Cmax | 18 months
Time to peak drug concentration-Tmax | 18 months
The area under the concentration-time curve from dosing (time 0) to time t-AUC0-t | 18 months
The time required for plasma concentration of a drug to decrease by 50%-t1/2 | 18 months
Treatment-related Adverse Event-TRAE | Until 28 days after the last dose of treatment

IPD SHARING:
Plan to Share IPD: No